CLINICAL TRIAL: NCT00765544
Title: Robot-assisted Ankle Rehabilitation for Multiple Sclerosis (Anklebot)
Brief Title: Targeted Lower Extremity Joint Training
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study re-design
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LO-0002
Record Dates: First submitted 2008-10-02; First posted 2008-10-03 (Estimated); Last update posted 2013-09-23 (Estimated); Status verified 2013-09

CONDITIONS: Multiple Sclerosis
Keywords: MS; Rehabilitation; Treadmill; Robot; Foot-drop
MeSH Terms: conditions — Multiple Sclerosis; Peroneal Neuropathies

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1 (Experimental): Anklebot
  Interventions: Device: Anklebot
- Arm 2 (Experimental): Body-weight supported treadmill training
  Interventions: Device: Lokomat
- Arm 3 (Experimental): Combination therapy (Anklebot and BWSTT)
  Interventions: Device: Anklebot; Device: Lokomat

INTERVENTIONS:
Device: Anklebot — The Ankle-Bot (Wheeler et al., 2004) is a stand-alone robot assisted device that is worn via a leather boot and knee brace (Fig.1). The Ankle-Bot can assist ankle movement throughout 3 planes. The percentage of force generated by the Ankle-Bot can be adjusted from no help, 0% assistance to 100% assistance. The device is low impedance and a subject can easily over come the forces generated by the Ankle-Bot. The Ankle-Bot will guide and assist the subject into ankle flexion, extension, inversion and eversion.
  Arms: Arm 1; Arm 3
Device: Lokomat — The Lokomat is a motor driven exoskeleton device that employs a body weight support suspension system and treadmill .
  Arms: Arm 2; Arm 3

SUMMARY:
The presence of foot drop limits normal gait. Our prior data has suggested that approximately 30% of MS patients have foot drop. Although we have observed that "task-specific" rehabilitation using the Lokomat can improve ambulation in chronic MS patients, subjects with "foot drop" have difficulty translating task-specific training to normative gait patterns over ground, despite improving speed and endurance.

One of the key limitations of the Lokomat is a lack of robot-assisted training for the ankle joint. The Anklebot, an MIT-developed rehabilitation robot for the ankle, has the potential to address this. The device can move throughout three planes and train ankle flexion, extension, inversion and eversion; however, therapy with the Anklebot alone does not train the knee or hip.

We plan to test whether subject foot drop and overall gait benefit more from Anklebot therapy alone or a combination of Anklebot and Lokomat.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of MS by McDonald criteria (McDonald, Compston et al. 2001). EDSS level between 3.5-5.5, who report ambulation problems.
2. Men and women between the ages 18-75 years.
3. Presence of unilateral foot drop that is clinically apparent to the PI or PI designate.
4. Must be able to ambulate 25 feet without an assisting device

Exclusion Criteria:

1. Cardiovascular: recent MI < 4 wk, uncontrolled HTN >190/110 mmHg, History of uncontrolled diabetes.
2. Symptoms of orthostasis when standing up.
3. Circulatory problems, history of vascular claudication or pitting edema.
4. Unable to fully understand instructions in order to use the equipment or the process of the study.
5. Body weight over 150 kg.
6. Lower extremity injuries that limit range of motion or function.
7. Joint problems (hip or leg) that limit range of motion or cause pain with movement despite treatment.
8. Unstable fractures.
9. Pressure sores with any skin breakdown in areas in contact with the body harness or Lokomat apparatus.
10. Chronic and ongoing alcohol or drug abuse.
11. Pre-morbid, ongoing depression or psychosis.
12. Ongoing physical therapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-09; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Strength and Gait | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Albert Lo, MD PhD, Principal Investigator — Providence VA Medical Center
Locations (1):
- Providence VA Medical Center, Providence, Rhode Island, United States